CLINICAL TRIAL: NCT05857150
Title: Exercise Response in Humans With Obesity
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian R. Lanza, Principal Investigator, Mayo Clinic
Other Study IDs: 22-012396
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obese
MeSH Terms: conditions — Obesity | interventions — Exercise Test; Absorptiometry, Photon; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample of DNA stored for possible future research use at Mayo Clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lean Group: Participants with body mass index 20-25 kg/m^2 will complete an outpatient study visit (body composition, blood draw, treadmill test, strength test) and an inpatient visit (muscle biopsies, fat biopsies, indirect calorimetry, exercise test).
  Interventions: Diagnostic Test: Treadmill Test; Diagnostic Test: Strength Test; Diagnostic Test: Dual-Energy X-Ray Absorptiometry; Procedure: Muscle Biopsy; Procedure: Fat Biopsy; Diagnostic Test: Resting Energy Expenditure; Diagnostic Test: Magnetic resonance imaging
- Obese Group: Participants with body mass index 30-45 kg/m^2 will complete an outpatient study visit (body composition, blood draw, treadmill test, strength test) and an inpatient visit (muscle biopsies, fat biopsies, indirect calorimetry, exercise test).
  Interventions: Diagnostic Test: Treadmill Test; Diagnostic Test: Strength Test; Diagnostic Test: Dual-Energy X-Ray Absorptiometry; Procedure: Muscle Biopsy; Procedure: Fat Biopsy; Diagnostic Test: Resting Energy Expenditure; Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Treadmill Test — Measurement of whole-body fitness level. Walking or running on a treadmill and breathing into a machine that measures oxygen level during test. Heart rhythm is continuously monitored during exercise using an electrocardiogram (ECG).
Diagnostic Test: Strength Test — Measure the strength of leg muscles by kicking against a machine with resistance.
Diagnostic Test: Dual-Energy X-Ray Absorptiometry — Body composition measurement.
  Other Names: DEXA
Procedure: Muscle Biopsy — Obtain a small piece of muscles from the upper part of the legs
Procedure: Fat Biopsy — Fat sample taken from abdomen
Diagnostic Test: Resting Energy Expenditure — Measured by indirect calorimetry. Measures how much energy the body uses at rest by placing a special plastic dome over the head while resting quietly for 30 minutes. Measures oxygen breathed in and carbon dioxide breathed out.
  Other Names: REE
Diagnostic Test: Magnetic resonance imaging — MRI on upper leg to look at fat and muscle
  Other Names: MRI

SUMMARY:
This study is being done to understand how chronic inflammation affects muscle function and responses to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Obese men and women ≥ 20 and ≤ 45 years of age.

Exclusion Criteria:

* Diabetes or fasting plasma glucose >126 mg/dL
* Anemia (female subjects hemoglobin of <11 g/dl and male subjects hemoglobin <12 g/dl)
* Active coronary artery disease or history of unstable macrovascular disease (unstable angina, myocardial infarction, stroke, and revascularization of coronary, peripheral or carotid artery within 3 months of recruitment)
* Renal failure (serum creatinine > 1.5mg/dl)
* Chronic active liver disease defined as aspartate aminotransferase (AST)>144 IU/L or alanine transaminase (ALT) >165 IU/L)
* Oral warfarin group medications or history of blood clotting disorders.
* Smoking
* Pregnancy or breastfeeding
* Alcohol consumption greater than 2 glasses/day or other substance abuse
* Untreated or uncontrolled hypothyroidism
* Debilitating chronic disease (at the discretion of the investigators)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men and women ages 20-45 years with Body Mass Index less than 25 or greater than 30 kg/m2.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change in muscle protein synthesis | Baseline, post-exercise approximately 8 hours
  Skeletal muscle protein synthesis will be measured from the rate of incorporation of infused amino acids measured by mass spectrometry.

SECONDARY OUTCOMES:
Change in mRNA expression of exercise responsive genes | Baseline, post-exercise approximately 8 hours
  Measure messenger ribonucleic acids (mRNAs) expression on exercise responsive genes
Change in expression and activation (phosphorylation) of signaling proteins | Baseline, post-exercise approximately 8 hours
  Phosphorylation is a common mechanism for the regulation of receptor function

CONTACTS AND LOCATIONS:
Overall Officials: Ian Lanza, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No